CLINICAL TRIAL: NCT00932542
Title: "Topic Effects of Eutectic Mixture Use in Local Anesthetics on Hemorrhoidectomy Postoperative (Prospective Study, Randomized, Triple Blind, Placebo-controlled)"
Brief Title: Eutectic Mixture for Hemorrhoidectomy Postoperative
Acronym: CRT054
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Collaborators: Cristália Produtos Químicos Farmacêuticos Ltda. (Industry)
Responsible Party: Principal Investigator, Joaquim Simoes Neto, Master Degree, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRT054
Record Dates: First submitted 2009-06-18; First posted 2009-07-03 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Hemorrhoidectomy
Keywords: Hemorrhoidectomy
MeSH Terms: interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Eutectic mixture (Experimental)
  Interventions: Drug: Eutectic mixture
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- Medicaina (Active Comparator)
  Interventions: Drug: lidocaine 2,5%; prilocaine 2,5%

INTERVENTIONS:
Drug: Eutectic mixture — The eutectic mixture of lidocaine + prilocaine + bupivacaine.
  Arms: Eutectic mixture
Drug: placebo — placebo
  Arms: placebo
Drug: lidocaine 2,5%; prilocaine 2,5% — lidocaine 2,5%; prilocaine 2,5%
  Arms: Medicaina

SUMMARY:
Assess the efficacy and safety of the topic use of an eutectic mixture of local anesthetics for postoperative pain control of patients submitted to hemorrhoidectomy. Patients will be operated and discharged at the same day in a day hospital clinic. During the fourteen days recovery period, they will apply the study medication to the anal region 4 times daily. The Visual Analog Pain Scale (VAS) will be answered twice daily. Patients will also take 100 mg oral nimesulide twice daily and 50 mg tramadol on demand up to 4 times daily. The tramadol demand will be tabulated. A rescue medication for analgesia will be provided (sodium diclofenac IM).

ELIGIBILITY:
Inclusion criteria: male and female patients, older than 18, having internal hemorrhoid disease grade III or IV with indication of elective surgery, anesthetic risk ASA 1 or 2; able to read and write.

Exclusion criteria: allergy or hypersensitivity to the mixture components, perianal fistulas, fissures, ulcers, infectious and inflammatory processes or tumors to the anal region, chronic diarrhea, megacolon or colonic anatomical deformities, hemorrhoidal thrombosis, gangrene or any condition that changes the indication from elective to urgent, previous surgery to anal-rectal region, history or clinical signs of diabetes mellitis type I or II, pregnancy, intense anxiety or important emotional disorder, participation in any clinical trial within the 3 months preceding the inclusion, investigator´s opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2010-04; Primary Completion 2011-02 (Actual); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Reduction of pain evaluated by the analgesics demand. | Follow-up termination (1 month)

SECONDARY OUTCOMES:
Pain reduction by VAS | Follow-up termination (1 month)
Tolerability by the adverse events incidence | Follow-up termination (1 month)

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Reis Neto, Campinas, São Paulo, Brazil